CLINICAL TRIAL: NCT05507008
Title: Starving for Energy - A Pilot Study to Test Ketone Derived Energy in Eating Disorders
Brief Title: Ketone Supplementation in Eating Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Guido Frank, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 804669
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa; Atypical Anorexia Nervosa; Atypical Bulimia Nervosa
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa

STUDY DESIGN:
Intervention Model Description: All subjects will complete 2-weeks daily ketone supplementation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketone Supplementation (Experimental): Subjects will ingest 2 daily doses of Kenetik ketone drink supplementation for 14 days.
  Interventions: Dietary Supplement: Kenetik Ketone Drink

INTERVENTIONS:
Dietary Supplement: Kenetik Ketone Drink — BHB supplementation

SUMMARY:
This study will investigate the effects of ketone supplementation on eating behavior including drive to binge eat or restrict, mood and anxiety in individuals with anorexia or bulimia nervosa. In addition, the investigators will contrast the effects of active ketone supplementation versus placebo on electroencephalogram (EEG) measurement. All subjects enrolled in the study will undergo EEG on two consecutive days at the beginning of the study, after active ketone supplementation or placebo drink, matched in taste to the ketone drink. Days will be randomized. Thereafter, all subjects will take the ketone supplementation drink for two weeks, twice daily.

DETAILED DESCRIPTION:
The goals of the study are:

1) to test the effect of BHB as a nutritional supplement for AN and BN and 2) to test the ingestion of BHB on brain function.

Subjects will complete a battery of self-assessments and a diagnostic assessment in order to determine eligibility and for characterization of behavior to be used in later analyses. After eligibility is confirmed, subjects will complete 2 EEG scans on separate days after ingestion of Ketone supplement drink or placebo and will complete a taste reward task during the EEG scan. Subjects will then complete 2 weeks of daily ketone supplementation and self-assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Must currently meet DSM-5 criteria for Anorexia Nervosa, Bulimia Nervosa, or OSFED Anorexia or Bulimia Nervosa based on the MINI diagnostic interview
2. Be medically stable as assessed by a comprehensive medical and behavioral evaluation conducted by a study physician
3. English as primary spoken language.
4. Ability to respond to EMA questions up to 6x per day within 60 minutes of receiving the message.

Exclusion Criteria:

1. Psychotic illness/other organic brain syndromes, dementia, somatization disorders or conversion disorders
2. Current substance abuse or dependence in the past 3 months
3. Physical conditions (e.g., diabetes mellitus, pregnancy) known to influence eating or weight
4. Medical conditions associated with ketoacidosis: type 1 diabetes mellitus, acute pancreatitis, alcoholic gastritis, peptic ulcer disease, hepatitis or Boerhaave syndrome (esophageal rupture)
5. History of significant head trauma
6. Indication of intellectual disability or autism spectrum disorder
7. Known allergy to any of the KenetikR drink components: D-beta-hydroxybutyric acid (D-BHB), Stevia, Monkfruit, Potassium Bicarbonate, Sodium Bicarbonate Potassium Sorbate or Taste Task Solutions: Sucrose, Potassium Chloride, Sodium bicarbonate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Eating Disorders Inventory 3 Drive for Thinness Subscale | Change from baseline to study completion, up to 2 weeks
  The Eating Disorders Inventory 3 is a self report assessment that measures core eating disorder symptoms. Subjects will complete this measure at the beginning and end of the study and the investigator will measure the change in scores. The Drive for Thinness Subscale has a range of 0 to 28 where higher scores mean worse outcome.
Eating Disorders Inventory 3 (EDI-3) Body Dissatisfaction Subscale | Change from baseline to study completion, up to 2 weeks
  The Eating Disorders Inventory 3 is a self report assessment that measures core eating disorder symptoms. Subjects will complete this measure at the beginning and end of the study and the investigator will measure the change in scores. The Drive for Thinness Subscale has a range of 0 to 40 where higher scores mean worse outcome.
Weight Change | Change in body mass index from baseline to study completion, up to 2 weeks]
  Body Mass Index over time as a measure of food intake from the start to end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Guido Frank, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mills IH, Park GR, Manara AR, Merriman RJ. Treatment of compulsive behaviour in eating disorders with intermittent ketamine infusions. QJM. 1998 Jul;91(7):493-503. doi: 10.1093/qjmed/91.7.493. PMID 9797933
- [Background] Frank GKW, Shott ME, Stoddard J, Swindle S, Pryor TL. Association of Brain Reward Response With Body Mass Index and Ventral Striatal-Hypothalamic Circuitry Among Young Women With Eating Disorders. JAMA Psychiatry. 2021 Oct 1;78(10):1123-1133. doi: 10.1001/jamapsychiatry.2021.1580. PMID 34190963
- [Background] Cheng B, Yang X, An L, Gao B, Liu X, Liu S. Ketogenic diet protects dopaminergic neurons against 6-OHDA neurotoxicity via up-regulating glutathione in a rat model of Parkinson's disease. Brain Res. 2009 Aug 25;1286:25-31. doi: 10.1016/j.brainres.2009.06.060. Epub 2009 Jun 25. PMID 19559687
- [Background] Kokkinou M, Ashok AH, Howes OD. The effects of ketamine on dopaminergic function: meta-analysis and review of the implications for neuropsychiatric disorders. Mol Psychiatry. 2018 Jan;23(1):59-69. doi: 10.1038/mp.2017.190. Epub 2017 Oct 3. PMID 28972576
- [Background] Brietzke E, Mansur RB, Subramaniapillai M, Balanza-Martinez V, Vinberg M, Gonzalez-Pinto A, Rosenblat JD, Ho R, McIntyre RS. Ketogenic diet as a metabolic therapy for mood disorders: Evidence and developments. Neurosci Biobehav Rev. 2018 Nov;94:11-16. doi: 10.1016/j.neubiorev.2018.07.020. Epub 2018 Jul 31. PMID 30075165